CLINICAL TRIAL: NCT01591499
Title: Clinical Evaluation of the Biofinity Multifocal Lens Compared With the Air Optix Aqua Multifocal Lens and With PureVision Multifocal Lens (INNOVATION PRESBYOPIA Study)
Brief Title: Clinical Evaluation of Biofinity Multifocal Compared With Air Optix Aqua Multifocal and With PureVision Multifocal
Acronym: INNOVATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-A00886-35
Record Dates: First submitted 2012-03-19; First posted 2012-05-04 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIOFINITY® MF - AIR OPTIX® AQUA MF (Experimental): During the first period, the participant will be allocated at random either the test lens pair (Biofinity) or a comparator lens pair (Air Optix or Purevision); during the second period, the participant will crossover to the alternate lens pair. (Biofinity crossover to Air Optix or Purevision) (Air Optix or Purevision crossover to Biofinity)
  Interventions: Device: BIOFINITY® MF - AIR OPTIX® AQUA MF; Device: BIOFINITY® MF - PUREVISION® MF
- BIOFINITY® MF - PUREVISION® MF (Active Comparator): During the first period, the participant will be allocated at random either the test lens pair (Biofinity) or a comparator lens pair (Air Optix or Purevision); during the second period, the participant will crossover to the alternate lens pair. (Biofinity crossover to Air Optix or Purevision) (Air Optix or Purevision crossover to Biofinity)
  Interventions: Device: BIOFINITY® MF - AIR OPTIX® AQUA MF; Device: BIOFINITY® MF - PUREVISION® MF

INTERVENTIONS:
Device: BIOFINITY® MF - AIR OPTIX® AQUA MF — During the first period, the participant will be allocated at random either the test lens pair (Biofinity) or a comparator lens pair (Air Optix or Purevision); during the second period, the participant will crossover to the alternate lens pair. (Biofinity crossover to Air Optix or Purevision) (Air Optix or Purevision crossover to Biofinity)
  Other Names: BIOFINITY® MULTIFOCAL; AIR OPTIX® AQUA MULTIFOCAL
Device: BIOFINITY® MF - PUREVISION® MF — During the first period, the participant will be allocated at random either the test lens pair (Biofinity) or a comparator lens pair (Air Optix or Purevision); during the second period, the participant will crossover to the alternate lens pair. (Biofinity crossover to Air Optix or Purevision) (Air Optix or Purevision crossover to Biofinity)
  Other Names: BIOFINITY® MULTIFOCAL; PUREVISION® MULTIFOCAL

SUMMARY:
This is a prospective, multi-centre, randomised, single-blind, cross-over study to compare the BIOFINITY® MULTIFOCAL lens and respectively the AIR OPTIX® AQUA MULTIFOCAL lens (lenses allocated on a ratio of 1/0.5) and the PUREVISION® MULTIFOCAL lens (lenses allocated on a ratio of 1/0.5), in presbyopic patients.

DETAILED DESCRIPTION:
This is a prospective, multi-centre, randomised, single-blind, cross-over study to compare the BIOFINITY® MULTIFOCAL lens and respectively the AIR OPTIX® AQUA MULTIFOCAL lens (lenses allocated on a ratio of 1/0.5) and the PUREVISION® MULTIFOCAL lens (lenses allocated on a ratio of 1/0.5), in presbyopic patients.

Each subject will have 5 visits with the investigator:

* (V1) An inclusion visit during which the first pair of lenses are fitted;
* (V2) An optimization visit after 7 to 9 days of wearing the first lens;
* (V3) An evaluation visit after an additional 10 to 15 days of wearing the first lens (17 to 24 days) and at which time the second pair of lenses are fitted;
* (V4, V5) Visits are conducted as in V 2 and V3 with the second pair of lenses.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, aged 18 years or older
* Patients with proven presbyopia
* Patients who do not wear contact lenses or who wore spherical lenses before being included in the study
* Myopic patients whose spherical equivalent is less than or equal to 9.00 D (or a "lens" power less than or equal to -8,00 D) or hypermetropic patients whose spherical equivalent is less than or equal to +5.50 D (or a "lens" power less than or equal to +6,00 D) or emmetropic patients for distance vision (plan)
* Patient able to fill in a diary without help
* Patients who gave their informed consent to take part in the study

Exclusion Criteria:

* Patients with a contra-indication for wearing contact lenses
* Patients suffering from any ocular pathology that might interfere with the evaluation of the lenses
* Patients wearing multifocal lenses or spherical lenses for monovision before being included in the study
* Astigmatic patients whose cylinder is more than 0.75 D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Cheneau, Study Director — CooperVision, Inc.; Caroline Bonneville, Study Director — CooperVision, Inc.; Catherine Peyre, Principal Investigator — Catherine Peyre

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multi-center study conducted by 15 freelance opthalmologiests to enroll 180 patients.
Groups:
- Biofinity Then Air Optix; Air Optix Then Biofinity; Biofinity Then Purevision; Purevision Then Biofinity: Randomized cross-over study to wear Biofinity Multifocal lenses or to wear either the Air Optix Aqual Multiocal lens (lenses allocated on a ratio of 1/0.5) or the PureVision Multifocal lens (lenses allocated on a ratio of 1/0.5).
  First pair of lens evaluated and worn up to 24 days. Subjects are crossed over to second pair of lens. Second pair of lens evaluated and worn up to 24 days.
Period: Baseline Visit
Arm/Group | Biofinity Then Air Optix | Air Optix Then Biofinity | Biofinity Then Purevision | Purevision Then Biofinity
Started | 33 | 39 | 31 | 39
Completed | 33 | 37 | 31 | 37
Not Completed | 0 | 2 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 2
Period: First Intervention (up to 24 Days)
Arm/Group | Biofinity Then Air Optix | Air Optix Then Biofinity | Biofinity Then Purevision | Purevision Then Biofinity
Started | 33 | 37 | 31 | 37
Completed | 33 | 37 | 31 | 37
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (up to 24 Days)
Arm/Group | Biofinity Then Air Optix | Air Optix Then Biofinity | Biofinity Then Purevision | Purevision Then Biofinity
Started | 33 | 37 | 31 | 37
Completed | 27 | 34 | 28 | 34
Not Completed | 6 | 3 | 3 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 0
Not completed — Lost to Follow-up | 4 | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Population of patients having evaluated at least one lens (N=132). Baseline characteristics was collected only for population having evaluated at least one lens.
Groups:
- Biofinity/Air Optix Aqua Combination: Participants were randomized to wear either a Biofinity pair or an Air Optix pair and then crossed over to the alternate lens pair. (Biofinity crossover to Air Optix or Air Optix crossover to Biofinity).
- Biofinity/Purevision Combination: Participants were randomized to wear either a Biofinity pair or an Purevision pair and then crossed over to the alternate lens pair. (Biofinity crossover to Purevision or Purevision crossover to Biofinity).
- Total: Total of all reporting groups
Arm/Group | Biofinity/Air Optix Aqua Combination | Biofinity/Purevision Combination | Total
Number analyzed (Participants) | 67 | 65 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] — Biofinity/Air Optix Combination - 3 missing values of subjects dispensed (N=70), Biofinity/Purevision Combination- 3 missing values of subjects dispensed (N=68).
  years | 53.51 (6.5) | 52.35 (5.48) | 52.94 (6.02)
Sex/Gender, Customized [Number; unit: participants] — Biofinity/Air Optix Combination (N=67, 3 missing values) Biofinity/Purevision Combination (N=66, 2 missing values)
  participants
    Female | 52 | 48 | 101
    Male | 15 | 17 | 32

OUTCOME MEASURES:

1. Secondary Outcome: Visual Performance - Near Visual Acuity
Description: Description: The participant's near binocular visual acuity (at 40 cm) using the Parinaud chart (smallest to largest letters, Score P1.5, P2, P4, P5) and reported per lens.
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 4 missing values; Air Optix Aqua Multifocal N=70, 8 missing values; Purevision Multifocal N=68, 8 missing values)
Measure: Number; unit: participants
Groups:
- Biofinity Multifocal: Visual performance by lens (Biofinity Multifocal) tested at V3 or V5
- Air Optix Aqua Multifocal: Visual performance by lens (Air Optix Aqua Multifocal)
- Purevision Multifocal: Visual performance by lens (Purevision Multifocal)
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 134 | 62 | 60
participants
  P1.5/P2 | 122 | 49 | 51
  P3 | 12 | 10 | 7
  P4 | 0 | 2 | 2
  P5 | 0 | 1 | 0

2. Primary Outcome: Visual Performance - Comparison of Initial Refraction to Multifocal Lenses
Description: The percentage of participants who obtained binocular distance and near visual acuities (VA) at least as good as their initial refraction assessment. Measured by Initial Refraction. Distance binocular VA (at 5 meters) using the Snellen chart decimal scale and near binocular VA (at 40 cm) using the Parinaud chart (smallest to largest letters, Score P1.5, P2, P4, P5).
  Change over time measured at V1 (initial refraction) and at V3 (lens pair one evaluation) and V5 (lens pair two evaluation):
  V1 = initial refraction at baseline, V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Change over time measured at V1, V3 and V5
Population: Percentage of patients who obtained distance and near binocular visual acuities at least as good as their initial refraction visual acuities.
  (Participant Flow: Biofinity Multifocal N=138, 14 missing values; Air Optix Aqua Multifocal N=70, 12 missing values; Purevision Multifocal N=68, 13 missing values)
Measure: Number; unit: percentage of participants
Groups:
- Biofinity Multifocal: Visual performance by lens (Biofinity Multifocal)
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 124 | 58 | 55
percentage of participants | 65.3 | 48.3 | 49.1

3. Secondary Outcome: Visual Performance - Distance Visual Acuity
Description: Description: The participant's distance binocular visual acuity (at 5 meters) using the La Galinet method. (Decimal scale, Excellent=between 5 and 20 tenths at 5 metres and between 1 and 20 tenths at 40 cm)
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measure at V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 5 missing values; Air Optix Aqua Multifocal N=70, 6 missing values; Purevision Multifocal N=68, 6 missing values)
Measure: Mean (Standard Deviation); unit: decimal units on a scale
Groups:
- Biofinity Multifocal: Visual performance by lens (Biofinity Multifocal) tested at visit V3 or V5
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 133 | 64 | 64
decimal units on a scale | 10.18 (1.51) | 9.87 (1.03) | 10.28 (1.3)

4. Secondary Outcome: Visual Performance - Quality of Near Vision
Description: Patients' subjective rating for quality of near vision by patient diary and reported per lens. (40cm away: reading a newspaper, looking at your watch etc. 0-100, 0=totally blurred, 100=perfectly clear).
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 3 missing values; Air Optix Aqua Multifocal N=70, 3 missing values; Purevision Multifocal N=68, 2 missing values)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 135 | 67 | 66
units on a scale | 83.19 (18.64) | 70.97 (26.3) | 71.27 (24.18)

5. Secondary Outcome: Visual Performance - Quality of Intermediate Vision
Description: Patients' subjective rating for quality of intermediate vision by patient diary and reported per lens. (distance equivalent to an arm's length. 0-100, 0=totally blurred, 100=perfectly clear).
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 3 missing values; Air Optix Aqua Multifocal N=70, 3 missing values; Purevision Multifocal N=68, 3 missing values)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 135 | 67 | 65
units on a scale | 81.25 (19.66) | 75.67 (23.56) | 76.08 (21.11)

6. Secondary Outcome: Visual Performance - Quality of Distance Vision
Description: Patients' subjective rating for quality of distance vision by patient diary and reported per lens. (driving, looking at a landscape, etc. 0-100, 0=totally blurred, 100=perfectly clear).
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at 17-24 days V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 4 missing values; Air Optix Aqua Multifocal N=70, 3 missing values; Purevision Multifocal N=68, 2 missing values)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 134 | 67 | 66
units on a scale | 73.54 (20.63) | 74.18 (20.75) | 74.33 (23.15)

7. Secondary Outcome: Visual Performance - Near, Low Contrast Vision
Description: The number of letters read at a near of 40 centimeters under 10% low contrast. Measured by objective assessment and reported per lens. Rated on a visual chart (La Galinet- number of letters read).
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 4 missing values; Air Optix Aqua Multifocal N=70, 4 missing values; Purevision Multifocal N=68, 4 missing values)
Measure: Mean (Standard Deviation); unit: number of letters read
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 134 | 66 | 64
number of letters read | 33.82 (11.74) | 31.76 (12.09) | 34.64 (12.07)

8. Secondary Outcome: Visual Performance: Near, High Contrast Vision
Description: The number of letters read at a near of 40 centimeters under 90% high contrast. Measured by objective assessment and reported per lens. Rated on a visual chart (La Galinet- number of letters read).
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at 17-24 days V3 or V5
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: number of letters read
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 134 | 66 | 64
number of letters read | 53.91 (12.72) | 49.11 (13.51) | 52.83 (12.8)

9. Secondary Outcome: Visual Performance: Distance, Low Contrast Vision
Description: The number of letters read at a distance of 5 meters under 10% low contrast. Measured by objective assessment and reported per lens. Rated on a visual chart (La Galinet- number of letters read).
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at V3 or V5
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: number of letters read
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 134 | 66 | 64
number of letters read | 19.09 (15.51) | 17.77 (15.43) | 18.77 (15.24)

10. Secondary Outcome: Visual Performance: Distance, High Contrast Vision
Description: The number of letters read at a distance of 5 meters under 90% high contrast. Measured by objective assessment and reported per lens. Rated on a visual chart (La Galinet- number of letters read).
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 5 missing values; Air Optix Aqua Multifocal N=70, 5 missing values; Purevision Multifocal N=68, 4 missing values)
Measure: Mean (Standard Deviation); unit: number of letters read
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 133 | 65 | 64
number of letters read | 39.76 (14.05) | 36.63 (14.71) | 38.75 (13.75)

11. Secondary Outcome: Visual Performance - Near Stereoscopic Vision
Description: The mean number of occurrences where the "number of the last figure where the patient equipped with analyzers can make out the raised circle (from number 1 to 9)," performed at a distance of 40 centimeters, using Wirt Vectographic Stereopsis Test. Reported per lens.
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 10 missing values; Air Optix Aqua Multifocal N=70, 7 missing values; Purevision Multifocal N=68, 4 missing values)
Measure: Mean (Standard Deviation); unit: number of occurrances
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 128 | 63 | 64
number of occurrances | 7.01 (2.38) | 6.21 (2.71) | 6.7 (2.69)

12. Secondary Outcome: Subjective Rating of Lens Comfort, Fitting
Description: Patients' subjective rating for lens comfort by patient diary and reported per lens. (After lens fitting, Scale 0-100, 0=very uncomfortable, 100=very comfortable).
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 7 missing values; Air Optix Aqua Multifocal N=70, 5 missing values; Purevision Multifocal N=68, 5 missing values)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Biofinity Multifocal: Comfort performance by lens (Biofinity Multifocal) tested at V3 or V5
- Air Optix Aqua Multifocal: Comfort performance by lens (Air Optix Aqua Multifocal)
- Purevision Multifocal: Comfort performance by lens (Purevision Multifocal)
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 131 | 65 | 63
units on a scale | 86.27 (17.65) | 80.77 (19.19) | 73.46 (24.26)

13. Secondary Outcome: Subjective Rating of Lens Comfort - During Day
Description: Patients' subjective rating for lens comfort by patient diary and reported per lens. (During the Day, Scale 0-100, 0=very uncomfortable, 100=very comfortable).
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 7 missing values; Air Optix Aqua Multifocal N=70, 5 missing values; Purevision Multifocal N=68, 4 missing values)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Biofinity Multifocal: Performance by lens (Biofinity Multifocal) tested at V3 or V5
- Air Optix Aqua Multifocal: Performance by lens (Air Optix Aqua Multifocal)
- Purevision Multifocal: Performance by lens (Purevision Multifocal)
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 131 | 65 | 64
units on a scale | 84.95 (16.63) | 81.54 (20.71) | 73.41 (23.4)

14. Secondary Outcome: Subjective Rating of Lens Comfort - End of Day
Description: Patients' subjective rating for lens comfort by patient diary and reported per lens. (At End of Day, Scale 0-100, 0=very uncomfortable, 100=very comfortable).
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at V3 or V5
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 131 | 65 | 63
units on a scale | 77.98 (20.66) | 73.51 (24.9) | 61.6 (27.78)

15. Secondary Outcome: Subjective Rating of Lens Comfort - General Comfort
Description: Patients' subjective rating for lens comfort by patient diary and reported per lens. (General Comfort, Scale 0-100, 0=very uncomfortable, 100=very comfortable).
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at V3 or V5
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 131 | 65 | 64
units on a scale | 85.66 (15.99) | 81.72 (21.51) | 70.75 (25.4)

16. Secondary Outcome: Comfort of Use - Average Wearing Time
Description: The average numbers of hours per day of lens wear by patient. Reported per lens. Calculated by number of hours worn.
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two Patients' subjective rating for lens comfort of use by patient diary and reported per lens. (Average Wearing Time in hours per day)
Time Frame: Measured at V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 11 missing values; Air Optix Aqua Multifocal N=70, 10 missing values; Purevision Multifocal N=68, 4 missing values)
Measure: Mean (Standard Deviation); unit: hours/day
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 127 | 60 | 62
hours/day | 11.61 (3.26) | 10.7 (3.04) | 11.27 (3.62)

17. Secondary Outcome: Geometric Performance - Lens Centration
Description: Description: The ophthalmologist's rating of lens centration during "Focus" and "Shift When Blinking" by questionnaire as a limited selected response (Optimal, Decentration Acceptable or Decentration Unacceptable). Assessed with the slit lamp and reported per lens.
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 12 missing values; Air Optix Aqua Multifocal N=70, 9 missing values; Purevision Multifocal N=68, 6 missing values)
Measure: Number; unit: Investigators
Groups:
- Biofinity Multifocal: Geometric performance by lens (Biofinity Multifocal) tested at V3 or V5
- Air Optix Aqua Multifocal: Geometric performance by lens (Air Optix Aqua Multifocal)
- Purevision Multifocal: Geometric performance by lens (Purevision Multifocal)
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 126 | 61 | 62
Investigators
  Optimal | 122 | 57 | 54
  Acceptable Shift | 4 | 4 | 8

18. Secondary Outcome: Geometric Performance - Lens Mobility
Description: The ophthalmologist's rating of lens movement during blinking by questionnaire as a limited selected response (Optimal, Acceptable with a tendency to be tight, Acceptable with a tendency to be Flat, Unacceptable and too tight, or Unacceptable too flat). Assessed with the slit-lamp and reported per lens.
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at 17-24 days V3 or V5
Population: (Participant Flow: Biofinity Multifocal N=138, 6 missing values; Air Optix Aqua Multifocal N=70, 5 missing values; Purevision Multifocal N=68, 5 missing values)
Measure: Number; unit: Investigators
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 132 | 65 | 63
Investigators
  Optimal | 116 | 58 | 49
  Acceptable Tight Tendency | 13 | 4 | 13
  Acceptable Flat Tendency | 3 | 3 | 1

19. Secondary Outcome: Clinical Performance - Lens Wettability
Description: The ophthalmologist's rating of lens wettability by questionnaire as a limited selected response (Zero, Low, Acceptable, Good or Excellent). Assessed with the slit lamp and reported per lens.
  Measured at V3 (lens pair one evaluation) or V5 (lens pair two evaluation):
  V3 = after 17-24 days of lens wear pair one, V5 = after 17-24 days of lens wear pair two
Time Frame: Measured at 17-24 days V3 or V5
Population: as for outcome 18
Measure: Number; unit: percentage of investigators
Groups:
- Biofinity Multifocal: Clinical performance by lens (Biofinity Multifocal) tested at V3 or V5
- Air Optix Aqua Multifocal: Clinical performance by lens (Air Optix Aqua Multifocal)
- Purevision Multifocal: Clinical performance by lens (Purevision Multifocal)
Arm/Group | Biofinity Multifocal | Air Optix Aqua Multifocal | Purevision Multifocal
Number analyzed (Participants) | 132 | 65 | 63
percentage of investigators
  None/Low/Acceptable | 31.1 | 53.8 | 52.4
  Good/Excellent | 68.9 | 46.2 | 47.6

20. Secondary Outcome: Lens Preference - Participant
Description: The number of participants who preferred a lens pair rated by diary questionnaire with a limited selected response.("Which pair of lenses did you prefer? The first pair, the second pair). Reported per lens.
  Measured at completion of V5 (lens pair two evaluation). Both lenses have been worn. Total time since base line is 34-48 days.
Time Frame: Measured at V5
Population: (Participant Flow: Biofinity Multifocal/Air Optix Aqua Multifocal N=70, 8 missing values; Biofinity Multifocal/Purevision Multifocal N=68, 7 missing values; Evaluated at least one lens N=138, 15 missing values.)
Measure: Number; unit: percentage of participants
Groups:
- Biofinity/Air Optix Combination: Participants were randomized to wear either a Biofinity pair or an Air Optix pair and then crossed over to the alternate lens pair. (Biofinity crossover to Air Optix) (Air Optix crossover to Biofinity)
- Biofinity/Purevision Combination: Participants were randomized to wear either a Biofinity pair or an Purevision pair and then crossed over to the alternate lens pair. (Biofinity crossover to Purevision) (Purevision crossover to Biofinity
- Evaluated At Least One Lens: Population of patients having evaluated at least one lens pair.
Arm/Group | Biofinity/Air Optix Combination | Biofinity/Purevision Combination | Evaluated At Least One Lens
Number analyzed (Participants) | 62 | 61 | 123
percentage of participants
  Biofinity | 59.7 | 77.0 | 68.3
  Air Optix | 40.3 | 0 | 20.3
  Purevision | 0 | 23.0 | 11.4

21. Secondary Outcome: Lens Preference - Ophthalmologist
Description: Ophthalmologists preference in terms of lenses rated by questionnaire with a limited selected response. ("Choice of Lens? First pair of lenses, Second pair of lenses") (Biofinity, Air Optix, or Purevision)
  Measured at completion of V5 (lens pair two evaluation). Both lenses have been worn. Total time since base line is 34-48 days.
Time Frame: Measured at 17-24 days V3 or V5
Population: (Participant Flow: Biofinity Multifocal/Air Optix Aqua Multifocal N=70, 8 missing values; Biofinity Multifocal/Purevision Multifocal N=68, 8 missing values; Evaluated at least one lens N=138, 16 missing values.)
Measure: Number; unit: percentage of investigators
Units Other Than Participants: lens Type
Arm/Group | Biofinity/Air Optix Combination | Biofinity/Purevision Combination | Evaluated At Least One Lens
Number analyzed (Participants) | 62 | 60 | 122
Number analyzed (lens Type) | 62 | 60 | 122
percentage of investigators
  Biofinity | 64.5 | 80.0 | 72.1
  Air Optix | 35.5 | 0 | 18.0
  Purevision | 0 | 20.0 | 9.8

ADVERSE EVENTS:
Time Frame: From dispense up to 24 days for both study lenses
Groups:
- Overall Study Population: Population of patients having evaluated at least one lens
Arm/Group | Overall Study Population
Serious Adverse Events (participants affected / at risk) | 0/138
Other Adverse Events (participants affected / at risk) | 0/138

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All the information collected during this study will be considered to be confidential until the analysis has been finalised by the study Sponsor.

All the data collected during this study will remain the property of the study Sponsor and may not be communicated to third parties under any circumstances without the Sponsor's express, written consent.

The results may not be published or passed on (orally or in writing) without the prior consent of the study sponsor.